CLINICAL TRIAL: NCT01679470
Title: A Pilot Study of AuroLase Therapy in Subjects With Primary and/or Metastatic Lung Tumors
Brief Title: Efficacy Study of AuroLase Therapy in Subjects With Primary and/or Metastatic Lung Tumors
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Nanospectra Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NBI-LC-001
Record Dates: First submitted 2012-08-13; First posted 2012-09-06 (Estimated); Last update posted 2016-11-03 (Estimated); Status verified 2016-11

CONDITIONS: Primary or Metastatic Lung Tumors
Keywords: cancer; lung; laser; ablation; airway obstruction
MeSH Terms: conditions — Lung Neoplasms; Neoplasms; Airway Obstruction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: AuroLase Therapy — Infusion of AuroShell particles followed by laser illumination for photothermal ablation of target lesions.

SUMMARY:
This is an open-label, single-center, single-dose efficacy pilot study of AuroLase Therapy in the treatment of subjects with primary and/or metastatic tumors of the lung where there is airway obstruction. In this study patients will be given a systemic IV infusion of particles and a subsequent escalating dose of laser radiation delivered by optical fiber via bronchoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have documented histological or cytological evidence of tumor(s) of the lung.
* Subjects must have one or more primary or metastatic tumors of the lung which have at least 10 mm in long axis as evaluated by spiral CT scan evaluation performed within last 30 days.
* Target lesions should be accessible to examination (examination by fiberoptic bronchoscopy is permitted) and to biopsy.
* Each index lesion should be large enough to provide at least 6 mg of tumor tissue by biopsy for assessment by neutron activation analysis.
* Tumors must be measurable according to RECIST criteria.
* Subjects must have ECOG Performance Score of 0, 1 or 2.
* Subjects must be ≥ 18 years of age.
* Subjects or their legal representative must be able to read, understand and sign an informed consent.
* Adequate renal function as evidenced by serum creatinine ≤ 2.0 mg/dL.
* Adequate hepatic function as evidenced by: Serum total bilirubin ≤ 2.0 mg/dL; Alkaline phosphatase ≤ 2X the ULN for the reference lab; SGOT/SGPT ≤ 2X the ULN for the reference lab.
* Women of childbearing potential must agree to use an effective form of contraception during the study and for 90 days following treatment (an effective form of contraception is an oral contraceptive or a double barrier method). Women who are NOT of childbearing potential are those who have undergone a bilateral oophorectomy or who have undergone menopause, defined as an absence of a menstrual cycle for 12 consecutive months.
* Negative pregnancy test for women of childbearing potential.

Exclusion Criteria:

* Subjects with known hypersensitivity to any of the components of the PEGylated AuroShell suspension (polyethylene glycol, gold).
* Patients who are pregnant and/or lactating.
* Patients who have undergone splenectomy.
* Subjects who are receiving concurrent investigational therapy or who have received investigational therapy within the 30 days prior to AuroShell infusion (investigational therapy is defined as treatment for which there is currently no regulatory authority approved indication).
* Subjects with evidence of an active bacterial infection or with a fever ≥ 38.5 ºC (101.3 ºF) within 3 days of the first scheduled day of dosing.
* Subject who has had a course of radiotherapy in the treatment area within the 30 days prior to AuroShell infusion.
* Subject who has had a course of chemotherapy or other anti-neoplastic therapy in the 30 days prior to AuroShell infusion.
* Life expectancy of less than 3 months.
* Any other medical condition, including mental illness or substance abuse, deemed by the Investigator to be likely to interfere with a subject's ability to sign informed consent, cooperate and participate in the study, or interfere with the interpretation of the results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2012-10; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Number of participants not manifesting a thermal lesion | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Glenn Goodrich, PhD, Study Director — Nanospectra Biosciences
Locations (1):
- Cancer Treatment Centers of America Eastern Regional Medical Center, Philadelphia, Pennsylvania, United States